CLINICAL TRIAL: NCT06293742
Title: A Phase 1, Open Label, Fixed Sequence Study to Evaluate the Effect of ECC5004 on the Single Dose Pharmacokinetics of Atorvastatin, Rosuvastatin, Digoxin and Midazolam in Healthy Participants
Brief Title: ECC5004 DDI Study With Atorvastatin, Rosuvastatin, Digoxin and Midazolam in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eccogene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EC0007
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Midazolam; Rosuvastatin Calcium; Digoxin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Digoxin, Rosuvastatin, ECC5004 (Part A) (Experimental): Part A consists of 2 treatment periods. Participants will receive Digoxin and Rosuvastatin administered alone in treatment period 1 and in combination with ECC5004 in treatment period 2.
  Interventions: Drug: ECC5004; Drug: Rosuvastatin; Drug: Digoxin
- Midazolam, Atorvastatin, ECC5004 (Part B) (Experimental): Part B consists of 5 treatment periods. In treatment period 1, participants will receive Midazolam administered alone followed by treatment period 2 in which participants will receive Atorvastatin administered alone. In treatment period 3, participants will receive ECC5004 alone. In treatment period 4, participants will receive ECC5004 in combination with Midazolam. In treatment period 5, ECC5004 will be administered alone and co-administered with Atorvastatin.
  Interventions: Drug: ECC5004; Drug: Midazolam; Drug: Atorvastatin
- Digoxin, Rosuvastatin, ECC5004 (optional Part C) (Experimental): Optional Part C consists of 2 treatment periods. Participants will receive Digoxin and Rosuvastatin administered alone in treatment period 1 and in combination with ECC5004 in treatment period 2.
  Interventions: Drug: ECC5004; Drug: Rosuvastatin; Drug: Digoxin
- Midazolam, Atorvastatin, ECC5004 (optional Part D) (Experimental): Optional Part D consists of 5 treatment periods. In treatment period 1, participants will receive Midazolam administered alone followed by treatment period 2 in which participants will receive Atorvastatin administered alone. In treatment period 3, participants will receive ECC5004 alone. In treatment period 4, participants will receive ECC5004 in combination with Midazolam. In treatment period 5, ECC5004 will be administered alone and co-administered with Atorvastatin.
  Interventions: Drug: ECC5004; Drug: Midazolam; Drug: Atorvastatin

INTERVENTIONS:
Drug: ECC5004 — ECC5004 tablet will be administered orally.
Drug: Midazolam — Midazolam will be administered orally.
  Arms: Midazolam, Atorvastatin, ECC5004 (Part B); Midazolam, Atorvastatin, ECC5004 (optional Part D)
Drug: Rosuvastatin — Rosuvastatin will be administered orally.
  Arms: Digoxin, Rosuvastatin, ECC5004 (Part A); Digoxin, Rosuvastatin, ECC5004 (optional Part C)
Drug: Digoxin — Digoxin will be administered orally.
  Arms: Digoxin, Rosuvastatin, ECC5004 (Part A); Digoxin, Rosuvastatin, ECC5004 (optional Part C)
Drug: Atorvastatin — Atorvastatin will be administered orally.
  Arms: Midazolam, Atorvastatin, ECC5004 (Part B); Midazolam, Atorvastatin, ECC5004 (optional Part D)

SUMMARY:
This is a Phase 1, open-label, non-randomized, fixed sequence study designed to evaluate the effect of ECC5004 on single dose pharmacokinetics of Atorvastatin, Rosuvastatin, Digoxin and Midazolam in healthy participants.

DETAILED DESCRIPTION:
The study consists of four parts (Part A, Part B, optional Part C and optional Part D), each with approximately 16 healthy participants enrolled. Part A and optional Part C of the study will have the same study design with two treatment periods, except that ECC5004 will be administered at a higher dose level in the optional Part C. Part B and optional Part D of the study will have the same study design with five treatment periods, except that ECC5004 will be administered at a higher dose level in optional Part D. Rosuvastatin and Digoxin will be administered alone or in combination with EC5004 in Part A and optional Part C. Atorvastatin and Midazolam will be administered alone or in combination with ECC5004 in Part B and optional Part D. The conduct of Part C and Part D with an increased dose of ECC5004 may be conducted as optional parts.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants of non-childbearing potential (NCBP) between the ages of 18 to 65 years of age
* BMI of 18.0 to 32.0 kg/m2
* Female participants who are postmenopausal, confirmed by FSH test, or surgically sterile, confirmed by medical documentation, or agree to practice true abstinence
* Male participants agree to use contraception, or agree to practice true abstinence
* No clinically significant findings in physical examination, 12-lead electrocardiogram (ECG), vital sign measurements, clinical laboratory evaluations, concomitant medications, or medical/psychiatric history
* Able to understand and sign and date informed consent

Exclusion Criteria:

* Females who are pregnant, planning to become pregnant, or breastfeeding during the study or within 3 months after the study
* Concomitant participation in any investigational study of any nature
* Blood loss of non-physiological reasons ≥ 200 ml (i.e., trauma, blood collection, blood donation) within 2 months prior to the first dose of study treatment, or plan to donate blood during this trial and within 1 month after the last dose of study treatment
* Serum calcitonin > 20 ng/L
* Clinically relevant acute or chronic medical conditions or diseases of the cardiovascular, gastrointestinal, hepatic, renal, endocrine, pulmonary, neurologic, psychiatric, immune or dermatologic systems
* Individual or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia 2 (MEN2), or suspected MTC
* History of pancreatitis
* Significant allergic reaction to active ingredients or excipients of the study drug
* Any clinically significant abnormal findings in the participant's physical examination, laboratory tests, pregnancy test, urine drug screen, alcohol test, or medical history which in the opinion of the Investigator would prevent the participants from participating in the study
* Used or plan to use any drugs or substances that can modulate the activity of CYP3A4 within at least 14 days prior to the first dose of study treatment until after their final follow up visit
* Use of drugs with enzyme-inducing properties such as St. John's Wort within 3 weeks prior to the first dose of study treatment until after their final follow up visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Atorvastatin PK parameters: AUC(0-tlast) | Part B and optional Part D: up to Day 34
  Area under the Plasma Concentration-Time Curve from Time 0 to the Last Measurable Non Zero Concentration
Atorvastatin PK parameters: AUC(0-inf) | Part B and optional Part D: up to Day 34
  Area under the Plasma Concentration-Time Curve from Time 0 Extrapolated to Infinity
Atorvastatin PK parameters: Cmax | Part B and optional Part D: up to Day 34
  Maximum observed plasma concentration
Rosuvastatin PK parameters: AUC(0-tlast) | Part A and optional Part C: up to Day 11
  Area under the Plasma Concentration-Time Curve from Time 0 to the Last Measurable Non Zero Concentration
Rosuvastatin PK parameters: AUC(0-inf) | Part A and optional Part C: up to Day 11
  Area under the Plasma Concentration-Time Curve from Time 0 Extrapolated to Infinity
Rosuvastatin PK parameters: Cmax | Part A and optional Part C: up to Day 11
  Maximum observed plasma concentration
Digoxin PK parameters: AUC(0-tlast) | Part A and optional Part C: up to Day 11
  Area under the Plasma Concentration-Time Curve from Time 0 to the Last Measurable Non Zero Concentration
Digoxin PK parameters: AUC(0-inf) | Part A and optional Part C: up to Day 11
  Area under the Plasma Concentration-Time Curve from Time 0 Extrapolated to Infinity
Digoxin PK parameters: Cmax | Part A and optional Part C: up to Day 11
  Maximum observed plasma concentration
Midazolam PK parameters: AUC(0-tlast) | Part B and optional Part D: up to Day 34
  Area under the Plasma Concentration-Time Curve from Time 0 to the Last Measurable Non Zero Concentration
Midazolam PK parameters: AUC(0-inf) | Part B and optional Part D: up to Day 34
  Area under the Plasma Concentration-Time Curve from Time 0 Extrapolated to Infinity
Midazolam PK parameters: Cmax | Part B and optional Part D: up to Day 34
  Maximum observed plasma concentration

SECONDARY OUTCOMES:
ECC5004 Safety parameters: Number of participants with adverse events (AEs) | Part A and optional Part C: up to Day 16; Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through adverse events
ECC5004 Safety parameters: Number of participants with vital sign abnormalities | Part A and optional Part C: up to Day 16; Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through vital signs
ECC5004 Safety parameters: Number of participants with electrocardiogram (ECG) abnormalities | Part A and optional Part C: up to Day 16; Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through electrocardiograms (ECGs)
ECC5004 Safety parameters: Number of participants with physical examination abnormalities | Part A and optional Part C: up to Day 16; Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through physical examination
ECC5004 Safety parameters: Number of participants with clinical laboratory abnormalities | Part A and optional Part C: up to Day 16; Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through clinical laboratory assessments
Atorvastatin safety parameters: Number of participants with adverse events (AEs) | Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through adverse events
Atorvastatin safety parameters: Number of participants with vital sign abnormalities | Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through vital signs
Atorvastatin safety parameters: Number of participants with electrocardiogram (ECG) | Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through electrocardiograms (ECGs)
Atorvastatin safety parameters: Number of participants with physical examination abnormalities | Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through physical examination
Atorvastatin safety parameters: Number of participants with clinical laboratory abnormalities | Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through clinical laboratory assessments
Rosuvastatin safety parameters: Number of participants with adverse events (AEs) | Part A and optional Part C: up to Day 16
  Safety Assessment evaluated through adverse events
Rosuvastatin safety parameters: Number of participants with vital sign abnormalities | Part A and optional Part C: up to Day 16
  Safety Assessment evaluated through vital signs
Rosuvastatin safety parameters: Number of participants with electrocardiogram (ECG) abnormalities | Part A and optional Part C: up to Day 16
  Safety Assessment evaluated through electrocardiograms (ECGs)
Rosuvastatin safety parameters: Number of participants with physical examination abnormalities | Part A and optional Part C: up to Day 16
  Safety Assessment evaluated through physical examination
Rosuvastatin safety parameters: Number of participants with clinical laboratory abnormalities | Part A and optional Part C: up to Day 16
  Safety Assessment evaluated through clinical laboratory assessments
Digoxin safety parameters: Number of participants with adverse events (AEs) | Part A and optional Part C: up to Day 16
  Safety Assessment evaluated through adverse events
Digoxin safety parameters: Number of participants with vital sign abnormalities | Part A and optional Part C: up to Day 16
  Safety Assessment evaluated through vital signs
Digoxin safety parameters: Number of participants with electrocardiogram (ECG) abnormalities | Part A and optional Part C: up to Day 16
  Safety Assessment evaluated through electrocardiograms (ECGs)
Digoxin safety parameters: Number of participants with physical examination abnormalities | Part A and optional Part C: up to Day 16
  Safety Assessment evaluated through physical examination
Digoxin safety parameters: Number of participants with clinical laboratory abnormalities | Part A and optional Part C: up to Day 16
  Safety Assessment evaluated through clinical laboratory assessments
Midazolam safety parameters: Number of participants with adverse events (AEs) | Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through adverse events
Midazolam safety parameters: Number of participants with vital sign abnormalities | Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through vital signs
Midazolam safety parameters: Number of participants with electrocardiogram (ECG) abnormalities | Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through electrocardiograms (ECGs)
Midazolam safety parameters: Number of participants with physical examination abnormalities | Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through physical examination
Midazolam safety parameters: Number of participants with clinical laboratory abnormalities | Part B and optional Part D: up to Day 40
  Safety Assessment evaluated through clinical laboratory assessments
ECC5004 PK parameters: AUC (0-τ) | Part A and optional Part C: up to Day 11; Part B and optional Part D: up to Day 34
  Area under the Plasma Concentration-Time Curve during the Dosing Interval
ECC5004 PK parameters: AUC(0-24) | Part A and optional Part C: up to Day 11; Part B and optional Part D: up to Day 34
  Area under the Plasma Concentration-Time Curve from Time 0 to 24 Hours Post-dose
ECC5004 PK parameters: tmax | Part A and optional Part C: up to Day 11; Part B and optional Part D: up to Day 34
  Time of the maximum observed plasma concentration
ECC5004 PK parameters: t1/2 | Part A and optional Part C: up to Day 11; Part B and optional Part D: up to Day 34
  Apparent terminal elimination half-life
ECC5004 PK parameters: CL/F | Part A and optional Part C: up to Day 11; Part B and optional Part D: up to Day 34
  Apparent Clearance
ECC5004 PK parameters: Ctau | Part A and optional Part C: up to Day 11; Part B and optional Part D: up to Day 34
  Observed Concentration at the End of the Dosing Interval

CONTACTS AND LOCATIONS:
Overall Officials: Eccogene, Study Director — Eccogene Clinical Trials
Locations (1):
- Eccogene Investigational Site, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No